CLINICAL TRIAL: NCT05683366
Title: Philps FAST picoSAT Pulse Oximetry Desaturation Study
Brief Title: Philps FAST2022 picoSAT Pulse Oximetry Desaturation Study
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: MA_PM_FAST 2022_2022_11492
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: SpO2 (Peripheral Oxygen Saturation) Measurement Validation
Keywords: Pulse Oximetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Group: No interventions, single group.
  Interventions: Device: No Intervention

INTERVENTIONS:
Device: No Intervention — There is no intervention in this study

SUMMARY:
Validation study to compare the accuracy of non-invasive Philips SpO2 sensors in detecting blood oxygen levels compared to invasive methods requiring a blood draw and lab analysis.

DETAILED DESCRIPTION:
To validate SpO2 accuracy performance of various SpO2 sensors with the Philips FAST Pulse Oximetry system during non-motion conditions over the range of 70-100% SaO2, arterial blood samples, assessed by CO-Oximetry

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent

  * Subject is 18 to 50 years of age
  * Subject must be willing and able to comply with study procedures and duration
  * Subject is a non-smoker or who has not smoked within 2 days prior to the study

Exclusion Criteria:

* Participant is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, wrist, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the particular sites utilized.) Female participants that are actively trying to get pregnant or are pregnant (confirmed by positive urine pregnancy test unless the participant is known to be not of child-bearing potential). Smoker Participants who have refrained will be screened for COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow) Participants with known respiratory conditions such as: (self-reported) uncontrolled / severe asthma flu pneumonia / bronchitis shortness of breath / respiratory distress unresolved respiratory or lung surgery with continued indications of health issues, emphysema, COPD, lung disease Participants with known heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review) hypertension: systolic >140mmHg, Diastolic >90mmHg on 3 consecutive readings (reviewed during health screen) have had cardiovascular surgery chest pain (angina) heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen) previous heart attack blocked artery unexplained shortness of breath congestive heart failure (CHF) history of stroke transient ischemic attack carotid artery disease myocardial ischemia myocardial infarction cardiomyopathy vascular diseases of the limbs Self-reported health conditions as identified in the Health Assessment Form (self-reported) diabetes, uncontrolled thyroid disease, kidney disease / chronic renal impairment, history of seizures (except childhood febrile seizures), epilepsy, history of unexplained syncope, recent history of frequent migraine headaches, recent symptomatic head injury (within the last 2 months) cancer / chemotherapy Self-reported dermatological conditions at application site severe dermatitis, hyperkeratosis (e.g., ichthyosis), nail fungus Participants with known clotting disorders (self-reported) history of bleeding disorders or personal history of prolonged bleeding from injury history of blood clots hemophilia current use of blood thinner: prescription or daily use of aspirin Sickle Cell Trait or Disease Participants with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported) Participants with severe allergies to iodine (only applicable if iodine is used) Participants with severe allergies to lidocaine (or similar pharmacological agents, e.g.

Novocaine) Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio < 0.4) Unwillingness or inability to remove colored nail polish from test digits. Dye injection within the past 48 hours Other known health condition, should be considered upon disclosure in health assessment form Dysfunctional hemoglobin levels

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population will include healthy non-smoking (or refrained from smoking for 2 days) competent adults, 18-50 yrs of age. It is planned that a sufficient number of participants will be screened to enroll in order to collect a minimum of 200 data points per sensor between 60 completed participants. Enrolled participants will be separated into 2 test groups of 30 completed participants. Each test group will consist of a minimum of 10 participants, with a min. of 3 males and 3 females, per each broad skin pigmentation category of light, medium, and dark.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Over 70-100% SpO2, an ARMS of ≤ 3.5% in non-motion conditions for the following SpO2 Sensor: 4053 | 13DEC2022-Q3 2023

SECONDARY OUTCOMES:
Over 70-100% SpO2, an ARMS of ≤ 3% in non-motion conditions for the following SpO2 Sensors: 989803128591, 989803205881, 989803205891, 989803205911, 989803205831, 989803205381, MAXAI, MAXNI, OxySoftN, 4004, and 4052 | 20DEC2022 - Q3 2023
  Over 70-100% SpO2, an ARMS of ≤ 2% in non-motion conditions for the following SpO2 Sensors: 989803144381, 989803205851, 4000, 4050, and 2258
  • Mean bias and limits of agreement for paired observations (SpO2 sensors and CO-Oximeter Over 70-100% SpO2, an ARMS within 1% among the broad categories of light, medium, and dark skin pigmentation for each SpO2 sensor under test Mean bias and limits of agreement for paired observations (SpO2 sensors and CO-Oximeter)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No